CLINICAL TRIAL: NCT05219123
Title: Inadvertent Pancreatic Duct Cannulation as an Independent Predictor of Post- Endoscopic Retrograde Cholangiopancreatography Pancreatitis
Brief Title: Guidewire Management in ERCP
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: McGill University (Other); University of Ottawa (Other); Queen's University (Other); Halton Health (Oakville) (Unknown); Island Health, Victoria, BC (Other)
Responsible Party: Sponsor
Other Study IDs: REB21-0940
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2022-01

CONDITIONS: ERCP
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No PD cannulation: Patients with native papilla undergoing ERCP for biliary indications with no inadvertent pancreatic duct cannulation
  Interventions: Other: ERCP with no PD cannulation
- Single PD cannulation: Patients with native papilla undergoing ERCP for biliary indications with a single inadvertent pancreatic duct cannulation with a guide wire
  Interventions: Other: ERCP with single PD cannulation

INTERVENTIONS:
Other: ERCP with no PD cannulation — ERCP with no PD cannulation
  Groups: No PD cannulation
Other: ERCP with single PD cannulation — ERCP with single PD cannulation
  Groups: Single PD cannulation

SUMMARY:
Intra-procedural guidewire management is a parameter whose impact remains incompletely understood in terms of its association with post- endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis (PEP). Inadvertent guidewire cannulation of the pancreatic duct (PD) when attempting common bile duct (CBD) cannulation is recognized as a risk factor for PEP. However, to date, no studies have assessed whether a single PD wire cannulation is associated with a higher PEP risk compared to no PD cannulations. Similarly, the relationship between each additional PD cannulation and the incremental magnitude of PEP risk remains unclear. In this study, the investigators will aim to assess whether a single inadvertent PD cannulation (versus no PD cannulation) is associated with an increased risk of PEP (the primary outcome).

DETAILED DESCRIPTION:
1. Background and Rationale

   While very effective, endoscopic retrograde cholangiopancreatography (ERCP) is widely known to have the highest adverse event (AE) profile among all commonly performed endoscopic procedures, with a collective AE rate of >10%. Common AEs include post-ERCP pancreatitis (PEP), bleeding, cholangitis, cholecystitis, perforation, and cardiopulmonary events. PEP is the most common, with estimated rates of 5-10%. It is noteworthy that both the incidence of PEP and its associated mortality are rising.

   It is of critical priority to patients, practitioners, and health administrators to investigate factors associated with all AEs and unplanned healthcare encounters (UHEs) following ERCP, especially given that most ERCPs are performed on an outpatient basis. The per-admission costs of post-ERCP UHEs are substantial, exceeding $10,000 and $70,000 for pancreatitis and cholangitis, respectively. PEP alone accounts for an estimated $200+ million in annual healthcare spending in the United States. Thus, researchers must prioritize the study of ERCP outcomes, striving to both identify and modify factors leading to AEs and UHEs.

   Intra-procedural guidewire management is a parameter whose impact remains incompletely understood. Inadvertent guidewire cannulation of the pancreatic duct (PD) when attempting common bile duct (CBD) cannulation is recognized as a risk factor for PEP. However, as inadvertent PD cannulation is highly correlated with difficult CBD cannulation in general, which itself is a risk factor for PEP, these associations are difficult to separate, even in randomized trials. To date, no studies have assessed whether a single PD wire cannulation is associated with a higher PEP risk compared to no PD cannulations. Similarly, the relationship between each additional PD cannulation and the incremental magnitude of PEP risk remains unclear.
2. Research Question and Objectives

   In this study, the investigators will aim to assess whether a single inadvertent PD cannulation (versus no PD cannulation) is associated with an increased risk of PEP (the primary outcome).
3. Methods

Design: Data will be used from the ongoing CReATE project (REB-18-0410). The exposure variable will be a single PD cannulation (versus no PD cannulation) in native papilla cases where the CBD was targeted for any indication. In addition to these variables, other parameters to be assessed include: the presence and timing of pharmacologic PEP prophylaxis, extent and timing of trainee involvement, the number and timing of common bile duct (CBD) cannulation attempts, the depth, timing, trajectory and number of PD cannulation(s), the presence and extent of PD opacification, the size(s) of sphincterotomy and/or sphincteroplasty, intra-procedural pathology, and the composition, caliber and length of any PD or CBD stent(s).

Outcomes: The primary outcome will be PEP, using established definitions. Secondary outcomes (defined a priori) will include PEP severity, overall and specific AEs (bleeding, cholangitis, cardio-pulmonary events), cannulation time and success rate, as well as overall procedure time and success rate.

Sample Size and Power: The investigators estimate 10,700 native papilla cases through the end of 2025. Extrapolating from our existing data (12.3% of eligible patients with a single PD cannulation and 69.4% with no PD cannulation), an estimated 1,316 patients will be exposed and an estimated 7,426 patients be controls. Assuming a two-sided alpha of 0.05, the investigators can demonstrate increases in PEP risk from 5.0% to 7.0% (a relative increase of 40%) with 82.1% power or from 5.0% to 7.5% (a relative increase of 50%) with 93.7% power.

Statistical Analysis: Variables will be compared using Student's t-test for measured variables and chi-squared test for categorical variables. P values < 0.05 will be considered significant. The investigators will use multivariable logistic regression to assess associations between risk factors and having PEP versus not having PEP. Clinically relevant subgroup analyses will also be performed by relevant patient-, endoscopist-, and procedure-related characteristics. Odds ratios per outcome will be reported with 95% CIs.

ELIGIBILITY:
Inclusion Criteria:

* Subject referred for ERCP, regardless of indication;
* Subject age 18 years or older;
* Subject able to give informed consent to involvement be included.

Exclusion Criteria:

* Previous sphincterotomy or sphincteroplasty
* Subject has a standard contraindication to ERCP;
* Subject or surrogate unable or unwilling to provide informed consent;
* Subject age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a hospital-based endoscopy unit for ERCP who have a native major papilla.
Sampling Method: Non-Probability Sample
Enrollment: 7461 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
post-ERCP pancreatitis | 30 days
  Defined using a previously published set of a priori criteria by indication (Cotton et al. Gastrointest Endoscopy 2010; 71:446-54).

CONTACTS AND LOCATIONS:
Overall Officials: Nauzer Forbes, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- Peter Lougheed Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No